CLINICAL TRIAL: NCT02811900
Title: An Evaluation of the Outcomes of Bariatric Surgery - a Cohort Study Internal Hernia After Laparoscopic Roux-en-Y Gastric Bypass: an Evaluation of the Impact on the Postoperative Course and a Quality of Life Case-control Study
Brief Title: An Evaluation of the Outcomes of Bariatric Surgery - a Cohort Study
Acronym: ChirBar
Status: Recruiting | Type: Observational
Sponsor: IHU Strasbourg (Other)
Responsible Party: Sponsor
Other Study IDs: 16-002-OBS
Record Dates: First submitted 2016-06-13; First posted 2016-06-23 (Estimated); Last update posted 2017-11-09 (Actual); Status verified 2017-11

CONDITIONS: Morbid Obesity
Keywords: obesity surgery; Roux en Y gastric bypass; sleeve gastrectomy; excess weight loss; quality of life
MeSH Terms: conditions — Obesity, Morbid | interventions — Gastric Bypass

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 30 Years
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: Roux en Y gastric bypass — Laparoscopic RYGB is performed as following: a gastric pouch of approximately 30mL was obtained using successive firings of the Endo GIATM linear stapler, followed by the creation of an antecolic alimentary limb of 150cm and of a biliopancreatic limb of 75cm. A gastrojejunal anastomosis was fashioned with the PCEEA™ 28 circular stapler until 2012, and using the Endo GIA™ linear stapler afterwards. The mesenteric defect and Petersen's defect were closed using a non-absorbable running suture.
Procedure: Sleeve gastrectomy — Laparoscopic SG is performed as following: after greater curvature mobilization, the gastric tube was calibrated over a 36F bougie and transection started approximately 5-6 cm from the pylorus toward the left diaphragmatic crus, using successive firings of 3.5- or 4.8-mm-high staples, depending on gastric thickness.
Procedure: Gastric banding — Laparoscopic gastric banding is performed as following: a perigastric tunel is performed by blunt dissection and the banding is calibrated over the stomach.
Procedure: Intragastric balloon — Flexible endoscopy is used to place intragastric balloon for a maximum interval of six months.

SUMMARY:
A prospective bariatric database was carried out in the Department of Digestive and Endocrine Surgery at the University Hospital of Strasbourg, France, starting in January 1996. All potential candidates for obesity surgery were prospectively registered in the database. Patients were informed by the bariatric surgeon of the prospective database, and of the possibility of utilizing personal data for research purpose after anonymization.

A case-control study was performed, to compare the quality of life (QoL) of patients treated for internal hernia (IH group) with the QoL of patients with an uncomplicated course after Roux en Y gastric bypass (Uncomplicated RYGB group).

DETAILED DESCRIPTION:
A prospective bariatric database was carried out in the Department of Digestive and Endocrine Surgery at the University Hospital of Strasbourg, France, starting in January 1996. All potential candidates for obesity surgery were prospectively registered in the database. Patients were informed by the bariatric surgeon of the prospective database, and of the possibility of utilizing personal data for research purpose after anonymization. Patients were evaluated by a multidisciplinary team. The standard preoperative assessment included nutritional counseling, psychological evaluation, abdominal ultrasound, upper gastrointestinal endoscopy, and blood tests. Type and date of surgery, biological and clinical follow-up data and morbidity data were recorded prospectively in the database.

A case-control study was performed, to compare the quality of life (QoL) of patients treated for internal hernia (IH group) with the QoL of patients with an uncomplicated course after Roux en Y gastric bypass (Uncomplicated RYGB group). Patients who had IH were paired with patients of the same age and sex and at the same postoperative interval. Paired patients were contacted by phone to obtain the QoL questionnaires, abdominal pain evaluation, and weight loss data.

ELIGIBILITY:
Inclusion Criteria:

* patient >18 years old
* BMI > 35 kg/m²

Exclusion Criteria:

* Incapacity of giving an informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient >18 years old BMI >35 kg/m²
Sampling Method: Non-Probability Sample
Enrollment: 10000 (Estimated)
Dates: Start 1996-01; Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Excess weight loss | 1 - 3 - 5 - 10 - 15 and 30 years

SECONDARY OUTCOMES:
BMI | 1 - 3 - 5 - 10 - 15 and 30 years
Albumin | 1 - 3 - 5 - 10 - 15 and 30 years
  Albumin
Pre-albumin | 1 - 3 - 5 - 10 - 15 and 30 years
  Pre-albumin
Vitamin A | 1 - 3 - 5 - 10 - 15 and 30 years
  Vitamin A
Vitamin D | 1 - 3 - 5 - 10 - 15 and 30 years
  Vitamin D
Vitamin B6 | 1 - 3 - 5 - 10 - 15 and 30 years
  Vitamin B6
Vitamin B9 | 1 - 3 - 5 - 10 - 15 and 30 years
  Vitamin B9
Vitamin B12 | 1 - 3 - 5 - 10 - 15 and 30 years
  Vitamin B12
Plasma ferritin | 1 - 3 - 5 - 10 - 15 and 30 years
  Plasma ferritin
Fasting plasma glucose | 1 - 3 - 5 - 10 - 15 and 30 years
  Fasting plasma glucose
Serum insulin | 1 - 3 - 5 - 10 - 15 and 30 years
  Serum insulin
HbA1c | 1 - 3 - 5 - 10 - 15 and 30 years
  HbA1c
Triglycerides | 1 - 3 - 5 - 10 - 15 and 30 years
  Triglycerides
Cholesterol | 1 - 3 - 5 - 10 - 15 and 30 years
  Cholesterol (total, HDL, LDL)
Quality of life assessed by Moorehead-Ardelt Quality of life II questionnaire | 1 - 3 - 5 - 10 - 15 and 30 years
  Moorehead-Ardelt Quality of life II questionnaire
Quality of life assessed by Gastro-intestinal Quality of Life Index | 1 - 3 - 5 - 10 - 15 and 30 years
  Gastro-intestinal Quality of Life Index
Postoperative morbidity | 1 - 3 - 5 - 10 - 15 and 30 years
  Postoperative morbidity

CONTACTS AND LOCATIONS:
Overall Officials: Didier Mutter, MD, PhD, Study Chair — Department of Digestive and Endocrine Surgery, University Hospital of Strasbourg
Locations (1):
- Service de Chirurgie Digestive et Endocrinienne, Strasbourg, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Lunca S, Vix M, Rikkers A, Rubino F, Marescaux J. Late gastric prolapse with pouch necrosis after laparoscopic adjustable gastric banding. Obes Surg. 2005 Apr;15(4):571-5. doi: 10.1381/0960892053723420. PMID 15946441
- [Result] Donatelli G, Costantino F, Dhumane P, Vix M, Perretta S, D' Agostino J, Dallemagne B, Marescaux J. Endoscopic intragastric balloon: a bridge toward definitive bariatric surgical management of a morbidly obese patient with situs ambiguous and midgut malrotation (with videos). Gastrointest Endosc. 2012 Jan;75(1):217-8. doi: 10.1016/j.gie.2011.01.022. Epub 2011 Mar 27. No abstract available. PMID 21444079
- [Result] Vix M, Diana M, Liu KH, D'Urso A, Mutter D, Wu HS, Marescaux J. Evolution of glycolipid profile after sleeve gastrectomy vs. Roux-en-Y gastric bypass: results of a prospective randomized clinical trial. Obes Surg. 2013 May;23(5):613-21. doi: 10.1007/s11695-012-0827-5. PMID 23207829
- [Result] Vix M, Liu KH, Diana M, D'Urso A, Mutter D, Marescaux J. Impact of Roux-en-Y gastric bypass versus sleeve gastrectomy on vitamin D metabolism: short-term results from a prospective randomized clinical trial. Surg Endosc. 2014 Mar;28(3):821-6. doi: 10.1007/s00464-013-3276-x. Epub 2013 Nov 7. PMID 24196556